CLINICAL TRIAL: NCT05080491
Title: Abnormal Thyroid Profile in Children With Attention Deficit With Hyperactivity Disorder (ADHD)
Brief Title: Thyroid Profile in Attention Deficit With Hyperactivity Disorder (ADHD)
Acronym: THYRADHD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fondation Lenval (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 21-HPNCL-04
Record Dates: First submitted 2021-09-30; First posted 2021-10-15 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2023-03

CONDITIONS: Attention Deficit With Hyperactivity Disorder
Keywords: ADHD; thyroid; free-T3; triiodothyronine; free-T4; thyroxine; TSH; chromatography; immuno-analysis; child; adolescent
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Thyroid Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Determination of thyroid profile and neuropsychological assessment (Experimental)
  Interventions: Diagnostic Test: immuno analysis and neuropsychological tests

INTERVENTIONS:
Diagnostic Test: immuno analysis and neuropsychological tests — A venous blood sample will be taken for assay in immuno-analysis including and for assay in chromatography with mass spectrometry. Patients will participate in computer neuropsychological tests: .
  Venous blood collection and the administration : the tubes are transported to the biochemistry laboratory of the University Hospital Center of Nice (CHU Nice) which prepares five aliquots (4 for assays in immuno-analysis including 2 on site, and one for assay in chromatography with mass spectrometry.
  Administration of two neuropsychological tests on computer(Attention Network Task and Tower of London).

SUMMARY:
Rationale: The observational data of University Children's Hospitals of Nice, suggest that about a quarter of children and adolescents with ADHD may present with an abnormal thyroid profile.

Main objective: To confirm that a subsample of children and adolescents with ADHD present with an abnormal thyroid profile using the gold standard for free fraction of hormones : chromatography with mass spectrometry.

Secondary objective: To examine to what extent this categorization holds using classic immuno-analytic assays. To characterize clinically and from a neuropsychological point of view this subsample and compare it to the other participants.

Study duration and design: 30 months (24 months for inclusion and 6 months for data analyses) open-label, (category 2 : interventional research with minimal risks or constraints), multicentre, without treatment or placebo administration.

Expected outcomes: Ancillary studies will investigate genetic physiopathological mechanisms (polymorphisms of deiodase or transmembrane carriers of thyroid hormones) and link this profile to other biological markers proposed in the literature (low ferritinemia, higher oxidative stress, atopic comorbid disease). The clinical trajectory of this subgroup and the persistence of this abnormal thyroid profile in adulthood will be a relevant issue in the future.

DETAILED DESCRIPTION:
Rationale: The internal observational data on 514 children and adolescents with ADHD suggest that 16-28% of them have an abnormal thyroid profile in immuno-analysis: normal free thyroid-stimulating hormone TSH and T4 but abnormally high free T3. Several pathophysiological hypotheses can be formulated, some of which relate to possible polymorphisms of the deiodase or transmembrane carriers of thyroid hormones, and also with other suspected biological markers of ADHD reported in the literature (low ferritin, atopic disease and oxidative stress). This abnormal thyroid profile may be an endophenotype of a subgroup of children and adolescents with ADHD. However, the reference technique for the determination of free fractions of hormones is chromatography with mass spectrometry and not immuno-analysis.

Main objective : To confirm by chromatography with mass spectrometry the existence of a subgroup of children and adolescents with ADHD with this abnormal thyroid profile.

Secondary objectives:

* Describe this subgroup by sex (male/female) and age (before 12 and after 12 years) clinically and neuropsychologically (Attention Network Task and Tower of London coupled with eye-tracking) and compare it with the rest of the sample.
* Dose thyroid hormones and TSH levels with 4 different techniques of immuno-analysis
* Calculate the classification concordance (abnormal profile / normal profile) between all pairs of dosage methods (chromatography and 4 immuno-analysis based techniques)
* Calculate 95% reference intervals for all assays and techniques throughout the sample.

Main evaluation criterion: free T3 greater than the 97.5 percentile of the reference interval in chromatography, free T4 between the 2.5 percentile and the 97.5 percentile with this same technique, and free TSH between the 2.5 percentile and the 97.5 percentile of the immuno-analytical reference interval.

Secondary evaluation criteria:

* Describe the subgroup and compare it to the rest of the sample:

  * Number of criteria for inattention, hyperactivity-impulsivity and therefore clinical presentation of ADHD (Predominant Inattentive, Predominant Hyperactive-Impulsive, Combined)
  * Scores for inattention, hyperactivity-impulsivity and their sum on the ADHD-Rating Scale and score on the Clinical Global Impression - Severity
  * Pattern of comorbidities diagnosed with Kiddie-SADDS-PL, manual, ocular and pedestrian preference, presence of atopic disease
  * Performance at the Attention Network Task and Test of the Tower of London coupled with eye-tracking
* Calculate the classification concordance all pairs of dosage methods (chromatography and 4 immuno-analysis based techniques): correlation, concordance indices 2x2 (for example, Cohen's kappa)
* Calculate 95% reference intervals with age as co-variable and separately for boys and girls.

Study duration: 30 months (24 months for inclusion and 6 months for data analyses) Study design: Open-label, cross-sectional (category 2 : interventional research with minimal risks or constraints), multicentre, no treatment or placebo administration.

Selection criteria:

* Inclusion criteria: Boys or girls aged 7 to 17 with ADHD (as per Diagnostic and Statistical Manual DSM-5 criteria).
* Criteria for Non-Inclusion:

  * Known or concurrent diagnosis of Autism Spectrum Disorder, Schizophrenia or Psychotic Disorder (as determined by DSM-5), thyroid disease of any origin, genetic disease known to affect thyroid function.
  * Any psychotropic treatment (for ADHD or others) in the month before inclusion or any treatment that may affect thyroid function
* Exclusion criteria: Withdrawal of informed consent by at least one of the child's parents or their legal representative.

Course of the study: The criteria for non-inclusion are checked, the diagnosis is confirmed using the Kiddie-SADS-PL before the child can be included. The patient's participation stops after the venous blood collection and the administration of two neuropsychological tests (Attention Network Task and Tower of London). The tubes are transported to the biochemistry laboratory of the CHU of Nice which prepares five aliquots (4 for assays in immuno-analysis including 2 on site, and one for assay in chromatography with mass spectrometry at the CHU of Toulouse).

Expected outcomes: The identification and clinical characterization of a subgroup of children and adolescents with ADHD with an abnormal thyroid profile will support the clinical diagnosis for these at least. Ancillary studies will investigate genetic physiopathological mechanisms (polymorphisms of deiodases or transmembrane carriers of thyroid hormones) and link this profile to other biological markers proposed in the literature (low ferritinemia, higher oxidative stress, atopic comorbid disease). The clinical trajectory of this subgroup and the persistence of this abnormal thyroid profile in adulthood will be relevant in the future

ELIGIBILITY:
Inclusion Criteria:

* Boys or girls aged by 7 and 17 years old included
* Diagnosed with ADHD according to DSM-5 criteria with either Inattentive predominant, Hyperactive-impulsive predominant or Combined presentations.
* Scoring at least 28 (maximum value 54) on the ADHD-RS total score that is the sum of 18 items each rated on a 0-3 scale.
* Scoring at least 4 (= Moderate) on the Clinical Global Impression - Severity scale
* Without any clinical symptom of either hypothyroidism or hyperthyroidism
* Who signed an informed consent form
* Whose at least of parents (or default a legal representative) signed an informed consent form

Exclusion Criteria:

Known or concomitant diagnosis of Autism Spectrum Disorder according to DSM-5 criteria Known or concomitant diagnosis of Schizophrenia or Psychotic Disorder according to DSM-5 criteria Known or concomitant diagnosis of any thyroid disorder (hypothyroidism or hyperthyroidism) whatever the cause might be Known or concomitant diagnosis of any genetic condition affecting the thyroid function (e.g. Down syndrome)

Intake in the last month of a psychotropic drug for:

ADHD: methylphenidate, atomoxetine, dexamphetamine, lisdexamphetamine, guanfacine or clonidine.

Any psychiatric disorder (antipsychotic, anxiolytics, antidepressant, etc.)

Intake in the last month of a molecule affecting the thyroid function:

* Any compound containing thyroid hormones
* Anti-thyroid drugs: carbimazole, thiamazole, propylthiouracil and perchlorate
* Any compound containing iodine
* Significant application on the skin of iodized products in the last six months
* Injection of water-soluble iodine contrast agents in the last 2 months or fat-soluble in the last 6 months

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 400 (Estimated)
Dates: Start 2023-11-21 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Definition of an abnormal thyroid profile | at inclusion
  To confirm by chromatography with mass spectrometry the existence of a subgroup of children and adolescents with ADHD with this abnormal thyroid profile. Free T3 greater than the 97.5 percentile of the reference interval in chromatography, free T4 between the 2.5 percentile and the 97.5 percentile with this same technique, and free TSH between the 2.5 percentile and the 97.5 percentile of the immuno-analytical reference interval.

SECONDARY OUTCOMES:
Describe the subgroup and compare it to pattern of comorbidities :ADHD Rating Scale | at inclusion
  measure of number of criteria for inattention, hyperactivity-impulsivity and therefore clinical presentation of ADHD (Predominant Inattentive, Predominant Hyperactive-Impulsive, Combined)
  ADHD Rating Scale: 9 inattention items and 9 hyperactivity-impulsivity items rated on a 0-3 scale (range 0-27), therefore the total score is on a 0-54 range. The higher the scores the higher the inattention and hyperactivity-impulsivity
Describe the subgroup and compare it to pattern of comorbidities :Kiddie-SADDS-PL | at inclusion
  measure of pattern of comorbidities diagnosed with Kiddie-SADDS-PL, manual, ocular and pedestrian preference, presence of atopic disease
  Kiddie-SADDS-PL: to make diagnoses according to DSM-V
Describe the subgroup and compare it to pattern of comorbidities: Performance at the Attention Network Task | at inclusion
  Determination of performance at the Attention Network Task (ANT) coupled with eye-tracking
  Three attention network will be assessed:
  Alerting: (RT without cue) minus (RT double cue) Orienting: (RT central cue) minus (RT orienting cue) Conflict: (RT flanker incongruent) minus (RT flanker congruent)
  Eye-tracking associated with ANT: On screen Areas Of Interest (AOI) are determined and for each of them the relative duration of gazing with be computed to build a patient-specific Task AOI : the fixation cross, cues and the target Peripheral AOI : the rest of the screen External AOI : outside the screen
Describe the subgroup and compare it to pattern of comorbidities: Performance at Tower of London | at inclusion
  Determination of performance at the test of the Tower of London coupled with eye-tracking.
  Tower of London: analysed variables are:
  Number of problems solved (maximum duration is one minute) Failure if three successive problems are unsolved Types of error : systematic rule violation, back-and-forth Percentage of problems solved with the execution (minimal) number of moves. Duration for planification and execution
Calculate the classification concordance all pairs of dosage methods | at inclusion
  Calculate the classification concordance (abnormal profile / normal profile) between all pairs of dosage methods (chromatography and 4 immuno-analysis based techniques)
Calculate 95% reference intervals with age as co-variable and separately for boys and girls. | at inclusion
  The age-dependent dosing curves with the reference interval for free-T3, free-T4 and TSH will be obtained by the method described by Royston et al. (1998) and Wright & Royston (1999).
Dose thyroid hormones and TSH levels with 4 different techniques of immuno-analysis | at inclusion
  Free-T3 and free-T4 dosed on different immuno-analyses techniques will be correlated

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpitaux Pédiatriques de Nice CHU-Lenval, Nice, France